CLINICAL TRIAL: NCT06071351
Title: Motivational Interviewing Based Training Program in Adults Effect on Reducing Cardiovascular Disease Risk Factors: A Randomized Controlled Trial
Brief Title: Motivational Interviewing Effect on Reducing Cardiovascular Disease Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Hasan EVCİMEN, Principal Investigator, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07/07/2023- 7/51
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Motivation; Nurse's Role; Risk Reduction
Keywords: cardiovascular disease; motivational interviewing; risk reduction; nurse's role
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention group (Experimental): In addition to the informative brochure prepared by the researcher, a 6-session motivational interview-based training program will be given. The training program will include topics such as nutrition, physical activity, smoking and alcohol use.
  Interventions: Other: motivational interviewing based training program
- Control Group (Active Comparator): An informative brochure prepared by the researcher and traditional consultancy services will be provided.
  Interventions: Other: Routine practice

INTERVENTIONS:
Other: motivational interviewing based training program — In addition to the informative brochure prepared by the researcher; A 6-session training program based on motivational interviewing, including nutrition, physical activity, smoking and alcohol use, will be held.
  Arms: Experimental intervention group
Other: Routine practice — An informative brochure prepared by the researcher was given.
  Arms: Control Group

SUMMARY:
Aim: The aim of this study is to examine the effect of motivational interviewing-based training program on reducing cardiovascular disease risk factors in adults.

Methods: In the first stage, individuals' CVD risk levels were determined. In the second stage, a 6-session motivational interview-based training program was applied to the intervention group with a medium CVD risk level (HearthSCORE score between 2 and 5 points). Brochures were distributed to the control group.

DETAILED DESCRIPTION:
The aim of this study is to determine the CVD risks of adult individuals between the ages of 40-70 and to evaluate the effect of a motivational interview-based training program on reducing modifiable risk factors in individuals with moderate CVD risk.

Hypothesis; A 6-session motivational interview-based training program aimed at reducing CVD risk factors reduces the risk level in the intervention group more than the control group.

This study will be carried out in 2 stages. In the first phase, risk prevalence screening will be carried out to determine the CVD risks of individuals between October and November 2023. In the 2nd phase, a randomized controlled study will be conducted to evaluate the intervention program for individuals at medium risk level (HeartScore® between 2 and 5).

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 40 and 70 years,
* Being voluntary to participate in the study,

Exclusion Criteria:

* Having a known and diagnosed CVD
* Not being voluntary to participate in the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-03-21 (Estimated)

PRIMARY OUTCOMES:
change is CVD risk level | 24 week
  In the first phase of the research, the "HeartScore®" program will be used to determine the CVD risk levels of individuals. Thanks to this program, the CVD risk levels of individuals will be learned and primary protection will be provided. According to "HeartScore®", CVD risk is discussed in 4 categories.
  * 10%, very high risk,
  * 5% - <10%, high risk, Medium risk between ≥2-<5%, If <1%, they are in the low risk category. As the score increases, the CVD risk level increases.

SECONDARY OUTCOMES:
Change in Physical Activity Level | 24 week
  Physical activity level was measured using the International Physical Activity Questionnaire Short Form (IPAQ).
  Sitting 1.5 MET Walking 3.3 MET Moderate Intensity Physical Activity 4.0 MET Vigorous Physical Activity 8.0 MET Short form (7 questions); It provides information on time spent awake, moderate to vigorous intensity activities, and time spent sitting. The IPAQ categorically classifies individuals as "inactive," "minimally active," and "very active."

CONTACTS AND LOCATIONS:
Locations (1):
- Kepez Devlet Hastanesi, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No